CLINICAL TRIAL: NCT01587963
Title: The Efficacy of High Dose Vitamin C in the Critically Ill Patient Population
Brief Title: High Dose Vitamin C in the Critically Ill Patient
Acronym: VitC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI's add. responsibilities and time commitment prevent him from completing trial
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 0220100048
Record Dates: First submitted 2012-04-26; First posted 2012-04-30 (Estimated); Results first posted 2017-05-11 (Actual); Last update posted 2017-05-11 (Actual); Status verified 2017-03

CONDITIONS: Shock
Keywords: hypovolemic or septic
MeSH Terms: conditions — Shock; Hypovolemia | interventions — Ascorbic Acid; Ringer's Lactate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ascorbic Acid (Active Comparator): Ascorbic Acid
  Interventions: Drug: Ascorbic Acid
- Ringers Lactate or Normal Saline (Placebo Comparator): Ringers Lactate or Normal Saline
  Interventions: Other: Ringers Lactate or Normal Saline

INTERVENTIONS:
Drug: Ascorbic Acid — 66mg/kg/hour of peripheral intravenous Vitamin C infusion for 24 hour duration, maximum total of 200 grams
  Other Names: Vit C
  Arms: Ascorbic Acid
Other: Ringers Lactate or Normal Saline — Fluid resuscitation will be given with NS or LR to achieve a same mean urine output of 0.5cc/kg/hour.
  Other Names: Placebo
  Arms: Ringers Lactate or Normal Saline

SUMMARY:
The purpose of this study is to determine the effectiveness of high doses of Vitamin C in critically ill patients.

DETAILED DESCRIPTION:
It has been shown that the stress that occurs during trauma, infection and/or shock depletes many of the body's resources such as Vitamin C (ascorbic acid) which may contribute to further complications. The purpose of this study is to determine the effectiveness of high doses of Vitamin C in critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* Activation of the Mass Transfusion Protocol following surgery or trauma.
* Diagnosis of septic shock. Septic shock will be defined as sepsis induced hypotension (i.e. systolic blood pressure <90mmHg or drop of systolic blood pressure >40mmHg in the presence of infection) that does not respond to a 2 liter fluid bolus.

Exclusion Criteria:

* Age less than 18 years.
* Pregnant women.
* Creatinine of greater than 2.2 g/dl at time of enrollment, history of chronic kidney or end stage renal disease, rise in creatinine > 1 g/dl within 24 hours prior to enrollment.
* Brain death diagnosed within 4 hours of presentation to the trauma bay or intensive care unit
* Patients with history of hemolytic blood disease, e.g. glucose-6-phosphate dehydrogenase deficiency, Sickle Cell Disease and Thalassemia.
* Patients in isolated cardiogenic shock.
* History of liver cirrhosis
* Transplant patients (liver, kidney, heart)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-02; Primary Completion 2014-02 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vicente Gracias, MD, Principal Investigator — RWJMS
Locations (1):
- Robert Wood Johnson University Hospital, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Ringers Lactate or Normal Saline
  Ringers Lactate or Normal Saline: Fluid resuscitation will be given with NS or LR to achieve a same mean urine output of 0.5cc/kg/hour.
Period: Overall Study
Arm/Group | Ascorbic Acid | Placebo
Started | 7 | 4
Completed | 6 | 4
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ascorbic Acid | Ringers Lactate or Normal Saline | Total
Number analyzed (Participants) | 7 | 4 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 3 | 9
  >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 4 | 1 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 7 | 3 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 5 | 4 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 4 | 11

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of High Dose Vitamin C Therapy in Shock Patients
Description: Given the grim prognosis of septic and hypovolemic shock, we aim to study the efficacy on an alternative treatment modality by implementing high dose vitamin C therapy in our patient population. Through previous investigations, especially research in the burn patient population, we expect that high dose vitamin C therapy will be beneficial to patients with hypovolemic or septic shock.
Time Frame: 30 days
Population: Study terminated prior to data collection completion. No data analysis performed.
Arm/Group | Ascorbic Acid | Ringers Lactate or Normal Saline
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Subjects will be randomized to receive high dose Vitamin C or placebo for 24 hours. The study team will follow the subjects and collect data through hospital discharge or 28 days whichever occurs first.
Arm/Group | Ascorbic Acid | Ringers Lactate or Normal Saline
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/4
Other Adverse Events (participants affected / at risk) | 0/7 | 0/4

LIMITATIONS AND CAVEATS:
Early termination leading to small number of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No